CLINICAL TRIAL: NCT06093828
Title: Transcatheter Treatment of Tricuspid Valve Regurgitation With the TriFlo Tricuspid Flow Optimizer (TFO) System
Brief Title: Transcatheter Treatment of Tricuspid Valve Regurgitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriFlo Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Symptomatic Severe Tricuspid Regurgitation

STUDY DESIGN:
Intervention Model Description: This study is a prospective single-arm, multicenter pre-market study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Other): Single-arm: subjects with Tricuspid valve regurgitation who meet the study eligibility criteria
  Interventions: Device: TriFlo Tricuspid Flow Optimizer

INTERVENTIONS:
Device: TriFlo Tricuspid Flow Optimizer — An introducer sheath is inserted into the femoral vein over a stiff guidewire; the sheath extends into the common iliac vein and inferior vena cava and in the right atrium. The TFO device is oriented coaxiality to the tricuspid. Once released, the delivery catheter and the steerable catheter are removed the access site closure performed by a cardiovascular or vascular surgeon or with pre-implanted percutaneous sutures per site preference.

SUMMARY:
Tricuspid Regurgitation induces an asymmetric enlargement of the tricuspid valve (TV) annulus causing a reduction of leaflets coaptation. Annular dilation continues even after surgical treatment. The progressive nature of TR, inadequate surgical treatment, and high-risk patient population make TR an ideal target for transcatheter therapy. The TriFlo TFO System introduces a new concept for the treatment of tricuspid regurgitation. Its commissural anchoring is designed to respect TV leaflet integrity, mobility, and maintain RV contractility.

DETAILED DESCRIPTION:
This study is a prospective single-arm, multicenter pre-market study. Recent epidemiological data estimate the prevalence of significant tricuspid regurgitation (TR) in the general population to be as high as 0.55% (and up to 3% after 75 years of age), a prevalence comparable to aortic stenosis (AS) or mitral regurgitation (MR). Although the prevalence is high, TR is often not treated. In the United States, approximately 1.6 million patients live with moderate to severe TR, and fewer than 8,000 tricuspid surgeries are performed annually.

Clinically relevant TR is present in approximately 3.0 million individuals in Europe and 70 million people worldwide. Approximately 90% of TR in adults is functional (secondary) and can be due to left-sided myocardial or valvular disease, pulmonary vascular disease, right ventricular myopathy,chronic right ventricular volume overload, or idiopathic. Uncertainty about the impact of TR on outcomes is related to the heterogeneous nature of the tricuspid disease, which is often secondary to other conditions (mainly left-sided disease or pulmonary hypertension). In spite of its high prevalence, tricuspid valve disease is a largely untreated condition and is known to be associated with poor life expectancy.

The purpose of this clinical study is to evaluate the safety and clinical efficacy of the TriFlo Tricuspid Flow Optimizer in the treatment of severe TR.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Symptomatic severe tricuspid regurgitation 3+ on a scale of 0+ to 5+, according to semi-quantitative echocardiographic color flow doppler evaluation
3. Tricuspid valve (TV) morphology which fulfills anatomic criteria of eligibility for the device according to Imaging Core Lab assessment
4. Signed (by subject or legal representative) and dated approved subject informed consent form prior to any study related procedure
5. Available and able to return to the study site for post-procedural follow-up examination

Exclusion Criteria:

CARDIOVASCULAR EXCLUSION CRITERIA

1. Requirement for an interventional percutaneous procedure or cardiac surgical procedure <30 days before or after index procedure
2. Prior tricuspid repair or replacement, implantation of an artificial heart valve.
3. Active endocarditis or history of endocarditis within the previous 12 months.
4. Left Ventricular Ejection Fraction <30%
5. Severe aortic and mitral stenosis and/or regurgitation
6. Severe tricuspid valve stenosis
7. Severe right ventricular failure
8. Systolic Pulmonary Artery pressure >70 mmHg
9. Echocardiographic evidence of intracardiac mass, thrombus, tumor, myxoma or vegetation
10. Femoral vein, inferior vena cava or evidence of intracardiac thrombus not adequately treated
11. Presence of an occluded or thrombosed inferior vena cava (IVC) filter that would interfere with the delivery catheter, or ipsilateral deep vein thrombosis is present.
12. Trans-tricuspid Pacemaker leads implanted within 90 days before the index procedure.

    EXCLUSION DUE TO COMORBIDITIES
13. Cerebrovascular event within the previous 6 months.
14. Myocardial infarction within 30 days prior to enrollment.
15. Bleeding disorders or hypercoagulable state, thrombocytopenia (platelet count <100,000/mm3), thrombocytosis (>750,000/mm3) or patient who refuses blood transfusions.
16. Acute anemia Hb<8 g/dl not adequately treated or white blood cell count<1000.
17. Severe renal failure requiring chronic dialysis or eGFR<25.
18. Severe Liver disfunction - class C cirrhosis.
19. Severe CLD with oxygen dependent COPD.
20. Coronary artery disease requiring revascularization

    EXCLUSION DUE TO CONTRAINDICATIONS
21. Unable to undergo transesophageal echocardiogram (TEE) and cardiac computed tomography (CT) or screening TEE is unsuccessful.
22. Contraindication, hypersensitivity or known allergy to device's components (nickel or titanium), aspirin, anti-coagulation and antiplatelet therapy or contrast media that cannot be adequately pre-medicated.
23. Known intolerance to anti-coagulation treatments.

    GENERAL EXCLUSION CRITERIA
24. Female patient pregnant (urine HCG test result positive) or lactating.
25. Known alcohol or drug abuser.
26. Currently participating in the study of an investigational drug or device.
27. Neoplasia with Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Acute safety, defined as freedom from device- or procedure-related Major Adverse Events (MAE) | 30 days
  a composite of death, Q-wave myocardial infarction, cardiac tamponade, cardiac surgery for failed TFO implantation, bleeding).

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Pineta Grande Hospital, Castel Volturno, Caserta
  - IRCCS Humanitas Research Hospital, Rozzano, Milano
  - IRCCS Policlinico San Donato, San Donato Milanese, Milano
  - Policlinico Campus Biomedico, Roma

IPD SHARING:
Plan to Share IPD: No